CLINICAL TRIAL: NCT03984617
Title: Impact of Football Matches on the Emergency Admissions of a Level III Maternity During EURO 2016
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS 2016/EURO-VIAL/ER
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Emergency visit in a French tertiary Maternity hospital (Maternity of Nancy) — total number of visits (hospitalizations and consultations)

SUMMARY:
Attendances at an emergency department (ED) are often considered to depend on different factors such as moonlight, welfare checks, weather, and major sporting events. Data regarding effects of large sporting events on the workload of ED often assessed decreased patient volume, especially male use. Currently, no data are available on the effect of major televised sporting events on obstetrical visits. The aim of this study is to examine whether televised soccer games from a major sporting tournament, (Euro 2016) influence the level of attendance at an obstetrical ED and could have implications for women's welfare.

In the summer of 2016, France hosted the largest European sporting event of the year 2016: the European Football Championships (Euro 2016). A total of 51 games were played over a month, bringing together the biggest European teams. An observational, retrospective study is conducted during this period on the number of emergency visits in a French tertiary Maternity hospital (Maternity of Nancy).

ELIGIBILITY:
Inclusion Criteria:

All female patients admitted urgently to the Regional Maternity Hospital between June 10 and July 10, 2016

Exclusion Criteria:

* refusal of the patient
* information and understanding impossible

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: All patients admitted to emergencies are informed of the protocol and a questionnaire is provided by the care team.
Sampling Method: Non-Probability Sample
Enrollment: 1114 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Overall number of maternity emergencies admissions during EURO 2016 (10June-10July) | At the end of EURO 2016 on 10th July 2016

SECONDARY OUTCOMES:
Number of daily admissions and per 2 hours time slot every day from June 10th to July 10th | At the end of EURO 2016 on 10th July 2016